CLINICAL TRIAL: NCT02836171
Title: Effect of Itraconazole on the Pharmacokinetics of Apatinib in Chinese Healthy Volunteers
Brief Title: Effect of Itraconazole on the Pharmacokinetics of Apatinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-APTN-DDI-03
Record Dates: First submitted 2016-07-14; First posted 2016-07-18 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2016-07

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — apatinib; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): subjects receiving a single 250 mg oral dose of apatinib mesylate tablets and wash-out for 3 days,then Itraconazole capsules 100 mg/day orally for 6 days with a single 250 mg oral dose of apatinib mesylate tablets co-administered on day 4 . apatinib mesylate tablets was administered in the morning after an overnight fast of at least 10 h
  Interventions: Drug: Apatinib Mesylate Tablets; Drug: Itraconazole Capsules

INTERVENTIONS:
Drug: Apatinib Mesylate Tablets — apatinib was administered in the morning after an overnight fast of at least 10 h
  Other Names: apatinib
Drug: Itraconazole Capsules — rifampicin was administered in the morning 0.5 hours after breakfast
  Other Names: itraconazole

SUMMARY:
he primary purpose of this study is to investigate potential pharmacokinetic interaction in healthy volunteers when apatinib is administered in combination with itraconazole. Secondary objective is evaluating the safety and tolerability of apatinib alone and when co-administered with itraconazole.

ELIGIBILITY:
Inclusion Criteria:

* female of non-childbearing potential or male;
* age 18-45 years;
* body mass index 19-24 kg/m2 with total body weight;

Exclusion Criteria:

* clinically signiWcant medical or surgical conditions with the potential to interfere with the absorption, distribution, metabolism or excretion of the study drugs;
* history of alcohol abuse; smoker;
* electrocardiogram(ECG) abnormality;
* blood pressure >140/90 mmHg;
* treatment with an investigational drug or any known CYP450 enzyme inducing/-inhibiting agents or herbal supplements within 14 days prior to first dose of study medication;
* Subjects were to abstain from using prescription and non-prescription drugs (other than acetaminophen as deemed necessary), vitamins and dietary supplements within 14 days prior to the first dose of study medication and throughout the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of Apatinib | 0~72h after apatinib administration

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From first administration to the seventh day after last administration
Peak Plasma Concentration (Cmax) of Apatinib | 0~72h after apatinib administration

CONTACTS AND LOCATIONS:
Overall Officials: Chen Yu, Principal Investigator — Shanghai Xuhui Central Hospital
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided